CLINICAL TRIAL: NCT03636217
Title: Effect of Kefir on Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zeynep Caferoglu, PhD, Assistant Professor Doctor, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: not defined
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Appetitive Behavior
Keywords: Appetite; Probiotic; Glycemic index
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LGI-Milk Breakfast (Experimental): Low glycemic index and milk content (LGI-Milk) breakfast as a test meal
  Interventions: Other: LGI-Milk Breakfast
- LGI-Kefir Breakfast (Experimental): Low glycemic index and kefir content (LGI-Kefir) breakfast as a test meal
  Interventions: Other: LGI-Kefir Breakfast
- HGI-Kefir Breakfast (Experimental): High glycemic index and kefir content (HGI-Kefir) breakfast as a test meal
  Interventions: Other: HGI-Kefir Breakfast

INTERVENTIONS:
Other: LGI-Milk Breakfast — This test meal with low glycemic index and milk were served as a breakfast after 12-hours fasting and participants were asked to consume the meal in full, within 15 min.
  Arms: LGI-Milk Breakfast
Other: LGI-Kefir Breakfast — In crossover design, this test meal with low glycemic index and kefir was served as a breakfast to compare the LGI-Milk Breakfast.
  Arms: LGI-Kefir Breakfast
Other: HGI-Kefir Breakfast — In crossover design, this test meal with high glycemic index and kefir was served as a breakfast to compare the LGI-Milk Breakfast and the LGI-Kefir Breakfast.
  Arms: HGI-Kefir Breakfast

SUMMARY:
This study aimed to determine the effect of kefir on appetite in healthy subjects. A randomized, single-blind, and 3-intervention crossover trial included 22 healthy and normal-weight (BMI 18.5-25 kg/m2) females aged 21-24 years. Participants were recruited to three test meals: an LGI-Milk, an LGI-Kefir, and an HGI-Kefir, with a one-week washout period. Appetite ratings were measured at 0, 15, 30, 60, 90, 120, 150, and 180 minutes. At the end of three hours, participants were served an ad libitum lunch meal. Then, the foods eaten at lunch were recorded and their energy and nutrient analysis was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal-weight (BMI 18.5-25 kg/m2)
* Female
* 21-24 years

Exclusion Criteria:

* During the last three months, change more than 5 kg in body weight or following an energy-restricted diet
* Being a vegan
* Having any chronic diseases such as diabetes, hypertension, etc.
* Physician-diagnosed medications or conditions that influence metabolism
* Smoking
* Practicing endurance sports
* Having difficulties with swallowing/eating
* Lack of appetite
* Hypersensitivity for the foods understudy
* Pregnant or lactating

Ages: 21 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Hunger rating | Three hours postprandial period
  Subjective assessment of appetite sensations was performed by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How hungry do you feel? (not at all hungry - as hungry as I ever felt)" at time points 0, 15, 30, 60, 90, 120, 150 and 180 minutes, and hunger rating was quantified as AUC (mm x min), which was calculated according to the trapezoidal rule by using those VAS scores. Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Fullness rating | Three hours postprandial period
  Subjective assessment of appetite sensations was performed by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How full do you feel? (not at all full - totally full)" at time points 0, 15, 30, 60, 90, 120, 150 and 180 minutes, and fullness rating was quantified as AUC (mm x min), which was calculated according to the trapezoidal rule by using those VAS scores. Total scale score changes in a range of 0-100. Higher values represent a better outcome.
Desiring to eat | Three hours postprandial period
  Subjective assessment of appetite sensations was performed by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How strong is your desire to eat? (very weak - very strong)" at time points 0, 15, 30, 60, 90, 120, 150 and 180 minutes, and desiring to eat was quantified as AUC (mm x min), which was calculated according to the trapezoidal rule by using those VAS scores. Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Prospective food consumption | Three hours postprandial period
  Subjective assessment of appetite sensations was performed by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How much do you think you can eat? (no food at all - a large amount of food)" at time points 0, 15, 30, 60, 90, 120, 150 and 180 minutes, and prospective food consumption was quantified as AUC (mm x min), which was calculated according to the trapezoidal rule by using those VAS scores. Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Composite appetite score | Three hours postprandial period
  The separate visual analog scale factors like hunger, fullness, desiring for eat, and prospective food consumption were combined to produce an additional measure termed 'composite appetite score'. This average appetite score was computed for 0, 15, 30, 60, 90, 120, 150 and 180 minutes using the following equation: [(hunger + desire to eat + prospective food consumption + (100 - fullness)]/4 Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Subsequent energy consumption | Three hours after the test breakfast
  Energy intake at ad libitum lunch was calculated.

SECONDARY OUTCOMES:
Desiring for sweet | Three hours postprandial period
  Subjective assessment of desire for specific food types was performed by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "Would you like to eat something sweet? (No, not at all - Yes, very much)" at time points 0, 15, 30, 60, 90, 120, 150 and 180 minutes, and desiring for sweet was quantified as AUC (mm x min), which was calculated according to the trapezoidal rule by using those VAS scores. Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Desiring for salty | Three hours postprandial period
  Subjective assessment of desire for specific food types was performed by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "Would you like to eat something salty? (No, not at all - Yes, very much)" at time points 0, 15, 30, 60, 90, 120, 150 and 180 minutes, and desiring for salty was quantified as AUC (mm x min), which was calculated according to the trapezoidal rule by using those VAS scores. Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Desiring for savoury | Three hours postprandial period
  Subjective assessment of desire for specific food types was performed by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "Would you like to eat something savoury? (No, not at all - Yes, very much)" at time points 0, 15, 30, 60, 90, 120, 150 and 180 minutes, and desiring for savoury was quantified as AUC (mm x min), which was calculated according to the trapezoidal rule by using those VAS scores. Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Desiring for fatty | Three hours postprandial period
  Subjective assessment of desire for specific food types was performed by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "Would you like to eat something fatty? (No, not at all - Yes, very much)" at time points 0, 15, 30, 60, 90, 120, 150 and 180 minutes, and desiring for fatty was quantified as AUC (mm x min), which was calculated according to the trapezoidal rule by using those VAS scores. Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Visual appeal of test meal | Immediately after consuming test meal (at 15 min)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How is the visual appeal of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Smell of test meal | Immediately after consuming test meal (at 15 min)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How is the smell of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Taste of test meal | Immediately after consuming test meal (at 15 min)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How is the taste of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Aftertaste of test meal | Immediately after consuming test meal (at 15 min)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "Is there any perceived taste in your mouth after test meal? (Much - None)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a better outcome.
Palatability of test meal | Immediately after consuming test meal (at 15 min)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How is the palatability of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Health Sciences, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03636217/Prot_SAP_001.pdf